CLINICAL TRIAL: NCT04677712
Title: MOBI: A Phase 4, Open-Label Study to Assess Effects of Mitigation Treatments on Bruising of CCH-aaes Treatment of Buttock Cellulite in Adult Females
Brief Title: Effects of Mitigation Treatments on Bruising of CCH-aaes Treatment of Buttock Cellulite
Acronym: MOBI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Collaborators: DeNova Research (Other); University of California, San Diego (Other); The Wall Center for Plastic Surgery (Other); Mathew Avram, MD (Unknown); Laser & Skin Surgery Medical Group, Inc. (Other); Investigate MD, LLC (Other); Biesman, Brian, M.D. (Individual); Plastic Surgical Associates of Fort Collins, P.C. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EN3835-401
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Edematous Fibrosclerotic Panniculopathy (EFP); Cellulite
Keywords: Bruising mitigation; CCH-aaes
MeSH Terms: conditions — Cellulite | interventions — Vascularin-Gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: CCH-aaes (Active Comparator): CCH-aaes was administered without mitigation treatment (control group).
  Interventions: Drug: CCH-aaes
- Cohort 2: CCH-aaes + Compression Garment (Active Comparator): CCH-aaes was administered with compression garment.
  Interventions: Other: Compression
- Cohort 3: CCH-aaes + Instant Cold Packs (Active Comparator): CCH-aaes was administered with instant cold packs.
  Interventions: Other: Cold Packs
- Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) (Active Comparator): CCH-aaes was administered with arnica gel patches (OcuMend).
  Interventions: Drug: Arnica Gel
- Cohort 5:CCH-aaes + INhance Post-Injection Serum with TriHex Technology® (Active Comparator): CCH-aaes was administered with INhance Post-Injection Serum with TriHex Technology®
  Interventions: Drug: INhance®
- Cohort 6: CCH-aaes + Pulse Dye Laser Treatment (PDL) (Active Comparator): CCH-aaes was administered with PDL.
  Interventions: Other: PDL

INTERVENTIONS:
Drug: CCH-aaes — Participants were administered CCH-aaes by subcutaneous injection to both buttocks.
  Other Names: QWO™
  Arms: Cohort 1: CCH-aaes
Other: Compression — Participants used a compression garment on both buttocks following subcutaneous CCH-aaes injections.
  Arms: Cohort 2: CCH-aaes + Compression Garment
Other: Cold Packs — Participants used cold packs applied to the right buttock for 5-10 minutes immediately after subcutaneous CCH-aaes injections.
  Arms: Cohort 3: CCH-aaes + Instant Cold Packs
Drug: Arnica Gel — Participants used Arnica Gel Patches (Arnica montana 50% and Ledum palustre) immediately after the CCH-aaes injection to the right buttock.
  Arms: Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend)
Drug: INhance® — Participants used INhance Post-injection Serum topically immediately after the CCH-aaes injection to the right buttock.
  Arms: Cohort 5:CCH-aaes + INhance Post-Injection Serum with TriHex Technology®
Other: PDL — Investigators applied one treatment with PDL to the right buttock between days 1-7 after injection.
  Arms: Cohort 6: CCH-aaes + Pulse Dye Laser Treatment (PDL)

SUMMARY:
This study will investigate treatments that may mitigate bruising after QWO™ (Collagenase clostridium histolyticum [CCH]-aaes) treatment of cellulite in the buttocks.

DETAILED DESCRIPTION:
CCH-aaes is indicated for the treatment of moderate to severe cellulite in the buttocks of adult women. Since bruising may be bothersome, this study will investigate treatments that may mitigate bruising after treatment of cellulite in the buttocks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have both buttocks with:

   1. Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS) score of 3 (moderate) as reported by the Investigator, and
   2. Hexsel Cellulite Severity Scale (CSS) Subsection D "Grade of laxity, flaccidity, or sagging skin" score of 0 (absence of laxity, flaccidity, or sagging skin) or 1 (slightly draped appearance).
2. Have a body mass index between ≥18 and ≤30 kilograms (kg)/square meter (m^2).
3. Be willing to apply sunscreen before each exposure to the sun while participating in the study (that is, Baseline through end of study).
4. Be judged to be in good health.
5. Be willing and able to cooperate with the requirements of the study.

Key Exclusion Criteria:

1. Has a coagulation disorder including but not limited to a Factor II, V, VII, or X deficiency.
2. Has local conditions in the areas to be treated (thrombosis, vascular disorder, active infection/inflammation, active cutaneous alteration, tattoo/mole) that restricts study participation.
3. Has skin laxity or linear undulations on buttocks that can be effaced by lifting skin.
4. Requires the following concomitant medications during the study and cannot discontinue these medications within the time specified before CCH-aaes treatment.

   1. Antiplatelet medication (clopidogrel [Plavix®] including aspirin at any dose within 14 days of treatment.
   2. Anticoagulants, such as warfarin (Coumadin®); heparin analogues within 14 days of treatment.
   3. Non-steroidal anti-inflammatory drugs (NSAIDS), such as ibuprofen (Motrin®, Advil®) and naproxen (Aleve®) 7 days before the study.
   4. Any medications or food that have or have been reported to have anticoagulant effects within 14 days of treatment.
   5. Antibiotics, such as penicillin and cephalosporin within 48 hours of treatment.
5. Has used or intends to use any of the local applications/therapies/injections/procedures that restricts study participation.
6. Is pregnant and/or is presently nursing or providing breast milk or plans to become pregnant during the study.
7. Intends to initiate an intensive sport or exercise program during the study.
8. Tanning or use of tanning agents.
9. Intends to engage in strenuous activity within 48 hours after the first injection of CCH-aaes.
10. Has received an investigational drug or treatment within 30 days prior to injection of CCH-aaes.
11. Has a history of hypersensitivity or allergy to collagenase or any other excipient of CCH-aaes.
12. Has a known systemic allergy or local sensitivity to any of the mitigation treatments or including excipients (that is, arnica patches, INhance Post-injection Serum).
13. Has received any collagenase treatments at any time prior to treatment in this study and/or has received EN3835 or CCH-aaes in a previous investigational study for cellulite.
14. For participants allocated to PDL treatment Participants will be excluded from PDL treatment if they have any contraindications to PDL a. exposure to Accutane® (isotretinoin) within 6 months of CCH-aaes treatment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Endo Pharmaceuticals
Locations (8):
- United States (8):
  - Endo Clinical Trial Site #3, Scottsdale, Arizona
  - Endo Clinical Trial Site #2, Sacramento, California
  - Endo Clinical Trial Site #7, San Diego, California
  - Endo Clinical Trial Site #6, Fort Collins, Colorado
  - Endo Clinical Trial Site #5, Chicago, Illinois
  - Endo Clinical Trial Site #1, Shreveport, Louisiana
  - Endo Clinical Trial Site #8, Boston, Massachusetts
  - Endo Clinical Trial Site #4, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: CCH-aaes: Collagenase clostridium histolyticum (CCH)-aaes was administered to both buttocks without mitigation treatment (control group).
- Cohort 2: CCH-aaes + Compression Garment: CCH-aaes was administered to both buttocks with compression garments as the mitigation treatment.
- Cohort 3: CCH-aaes + Instant Cold Packs: CCH-aaes was administered to both buttocks with instant cold packs applied to the right buttock only for 5-10 minutes post injection as the mitigation treatment.
- Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend): CCH-aaes was administered to both buttocks with arnica gel patches (OcuMend) applied to the right buttock only immediately after injection and twice daily (BID) for 2 days as the mitigation treatment.
- Cohort 5: CCH-aaes + INhance Post-Injection Serum With TriHex Technology®: CCH-aaes was administered to both buttocks with INhance Post-Injection Serum with TriHex Technology® applied to the right buttock only four times daily (QID) for up to 7 days as the mitigation treatment.
- Cohort 6: CCH-aaes + Pulse Dye Laser Treatment (PDL): CCH-aaes was administered to both buttocks with PDL applied once to the right buttock only between Days 1-7 post injection as the mitigation treatment.
Period: Overall Study
Arm/Group | Cohort 1: CCH-aaes | Cohort 2: CCH-aaes + Compression Garment | Cohort 3: CCH-aaes + Instant Cold Packs | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) | Cohort 5: CCH-aaes + INhance Post-Injection Serum With TriHex Technology® | Cohort 6: CCH-aaes + Pulse Dye Laser Treatment (PDL)
Started | 7 | 8 | 9 | 9 | 8 | 7
Received at Least 1 Dose of Study Drug | 7 | 8 | 9 | 9 | 8 | 7
Completed | 7 | 7 | 9 | 9 | 8 | 7
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants allocated to treatment who received at least 1 injection of CCH-aaes with or without mitigation treatment
Groups:
- Cohort 1: CCH-aaes: CCH-aaes was administered to both buttocks without mitigation treatment (control group).
- Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend): CCH-aaes was administered to both buttocks with arnica gel patches (OcuMend) applied to the right buttock only immediately after injection and BID for 2 days as the mitigation treatment.
- Cohort 5:CCH-aaes + INhance Post-Injection Serum With TriHex Technology®: CCH-aaes was administered to both buttocks with INhance Post-Injection Serum with TriHex Technology® applied to the right buttock only QID for up to 7 days as the mitigation treatment.
- Cohort 6: CCH-aaes + PDL: CCH-aaes was administered to both buttocks with PDL applied once to the right buttock only between Days 1-7 post injection as the mitigation treatment.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: CCH-aaes | Cohort 2: CCH-aaes + Compression Garment | Cohort 3: CCH-aaes + Instant Cold Packs | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) | Cohort 5:CCH-aaes + INhance Post-Injection Serum With TriHex Technology® | Cohort 6: CCH-aaes + PDL | Total
Number analyzed (Participants) | 7 | 8 | 9 | 9 | 8 | 7 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (6.32) | 37.8 (9.06) | 38.4 (6.85) | 37.8 (7.37) | 41.4 (8.01) | 39.4 (5.88) | 39.0 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 9 | 9 | 8 | 7 | 48
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 1 | 2 | 6
  Not Hispanic or Latino | 5 | 8 | 9 | 8 | 7 | 5 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 7 | 7 | 9 | 9 | 8 | 7 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.46 (3.182) | 26.54 (2.729) | 24.68 (3.440) | 25.50 (3.094) | 26.81 (2.645) | 24.97 (2.759) | 25.51 (2.978)
Fitzpatrick Skin Rating [Number; unit: units on a scale]
  I (Pale White) | 0 | 2 | 0 | 1 | 0 | 0 | 3
  II (Fair) | 3 | 2 | 5 | 4 | 5 | 3 | 22
  III (Darker White) | 4 | 4 | 4 | 4 | 3 | 4 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants by Buttock at Each Level of Bruising on the Investigator Assessment of Bruising Severity Scale at Day 4
Description: Participants were assessed by the investigator using the Investigator Assessment of Bruising Severity Scale. The Investigator Assessment of Bruising Severity Scale is a 5-point photonumeric scale ranging from 0 to 4, with "0" indicating no bruising or almost none, and "4" indicating very severe bruising. Higher scores indicated worse outcome.
Time Frame: Day 4 (3 days after CCH-aaes injection)
Population: Evaluable Population: All participants allocated to treatment who receive at least 1 injection of CCH-aaes and had at least 1 bruising assessment after the first dose of CCH-aaes.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 5: CCH-aaes + Post-Injection Serum With TriHex Technology®: CCH-aaes was administered to both buttocks with INhance Post-Injection Serum with TriHex Technology® applied to the right buttock only QID for up to 7 days as the mitigation treatment.
Arm/Group | Cohort 1: CCH-aaes | Cohort 2: CCH-aaes + Compression Garment | Cohort 3: CCH-aaes + Instant Cold Packs | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) | Cohort 5: CCH-aaes + Post-Injection Serum With TriHex Technology® | Cohort 6: CCH-aaes + PDL
Number analyzed (Participants) | 7 | 8 | 9 | 9 | 8 | 7
Participants
  Left Buttock (control): None or almost no bruising (0) | 0 | 0 | 0 | 0 | 0 | 0
  Right Buttock: None or almost no bruising (0) | 0 | 0 | 0 | 0 | 0 | 0
  Left Buttock (control): mild bruising (1) | 2 | 2 | 5 | 1 | 1 | 3
  Right Buttock: mild bruising (1) | 2 | 3 | 5 | 1 | 1 | 4
  Left Buttock (control): Moderate bruising (2) | 1 | 3 | 3 | 3 | 2 | 2
  Right Buttock: Moderate bruising (2) | 1 | 2 | 3 | 4 | 3 | 2
  Left Buttock (control): severe bruising (3) | 3 | 3 | 1 | 4 | 5 | 1
  Right Buttock: severe bruising (3) | 3 | 3 | 1 | 3 | 4 | 1
  Left Buttock (control): very severe bruising (4) | 1 | 0 | 0 | 1 | 0 | 1
  Right Buttock: severe bruising (4) | 1 | 0 | 0 | 1 | 0 | 0

2. Secondary Outcome: Number of Participants for Whom The Investigator Reported an Improvement of Bruising on the Mitigation-treated Buttock as Measured on the Investigator-Bruising Improvement Scores (I-BIS)
Description: The investigator assessed improvement of bruising using the I-BIS, a 3-point Likert scale that compares bruising on the mitigated side to the bruising on the non-mitigated side as either worse (1), the same (2), or improved (3). I-BIS Rating was directly obtained from the investigator's assessment rating comparing the bruising of the mitigation-treated buttock to the untreated (with mitigation treatment) buttock.
Time Frame: Days 4 and 7
Population: Evaluable Population: All participants allocated to treatment who received at least 1 injection of CCH-aaes and had at least 1 bruising assessment after the first dose of CCH-aaes. The I-BIS assessment was not completed for participants that did not receive mitigation treatment (Cohort 1) or participants that received bilateral mitigation treatment (Cohort 2), as these participants did not have an untreated buttock as a comparator.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: CCH-aaes + Instant Cold Packs | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) | Cohort 5:CCH-aaes + INhance Post-Injection Serum With TriHex Technology® | Cohort 6: CCH-aaes + PDL
Number analyzed (Participants) | 9 | 9 | 8 | 7
Participants
  Day 4 | 2 | 4 | 2 | 4
  Day 7 | 4 | 5 | 5 | 4

3. Secondary Outcome: Number of Participants With an Improvement of Bruising on the Mitigation Treated Buttock on the Subject-Bruising Improvement Scale (S-BIS)
Description: The investigator assessed improvement of bruising using the S-BIS, a 3-point Likert scale that compares bruising on the mitigated side to the bruising on the non-mitigated side as either worse (1), the same (2), or improved (3). S-BIS Rating was directly obtained from the participant's assessment rating comparing the bruising of the mitigation-treated buttock to the untreated (with mitigation treatment) buttock. The S-BIS assessment was not completed for participants that did not receive mitigation treatment (Cohort 1) or participants that received bilateral mitigation treatment (Cohort 2), as these participants did not have an untreated buttock as a comparator.
Time Frame: Days 4 and 7
Population: Evaluable Population: All participants allocated to treatment who received at least 1 injection of CCH-aaes and had at least 1 bruising assessment after the first dose of CCH-aaes. The S-BIS assessment was not completed for participants that did not receive mitigation treatment (Cohort 1) or participants that received bilateral mitigation treatment (Cohort 2), as these participants did not have an untreated buttock as a comparator.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 5: CCH-aaes + INhance Post-Injection Serum With TriHex Technology®: CCH-aaes was administered to both buttocks with INhance Post-Injection Serum with TriHex Technology® applied to the right buttock only QID for up to 7 days as the mitigation treatment.
Arm/Group | Cohort 3: CCH-aaes + Instant Cold Packs | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) | Cohort 5: CCH-aaes + INhance Post-Injection Serum With TriHex Technology® | Cohort 6: CCH-aaes + PDL
Number analyzed (Participants) | 9 | 9 | 8 | 7
Participants
  Day 4 | 0 | 3 | 1 | 3
  Day 7 | 4 | 4 | 3 | 4

4. Secondary Outcome: Number of Participants Bothered by the Appearance of Bruising as Assessed by the Patient Bother by Bruising Scale at Day 4
Description: The Patient Bother by Bruising Scale is a 4-point scale, with a score of 1 indicating not bothered at all, and a score of 4, indicating extremely bothered. A lower score indicates a better outcome.
Time Frame: Day 4
Population: Evaluable Population: All participants allocated to treatment who received at least 1 injection of CCH-aaes and had at least 1 bruising assessment after the first dose of CCH-aaes.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: CCH-aaes | Cohort 2: CCH-aaes + Compression Garment | Cohort 3: CCH-aaes + Instant Cold Packs | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) | Cohort 5: CCH-aaes + INhance Post-Injection Serum With TriHex Technology® | Cohort 6: CCH-aaes + PDL
Number analyzed (Participants) | 7 | 8 | 9 | 9 | 8 | 7
Participants
  Left Buttock (control): Not at all bothered (1) | 3 | 5 | 9 | 5 | 4 | 1
  Right Buttock: Not at all bothered (1) | 3 | 5 | 9 | 5 | 4 | 1
  Left Buttock (control): A little bothered (2) | 3 | 2 | 0 | 2 | 2 | 4
  Right Buttock: A little bothered (2) | 3 | 2 | 0 | 2 | 2 | 4
  Left Buttock (control): Moderately bothered (3) | 1 | 1 | 0 | 2 | 2 | 1
  Right Buttock: Moderately bothered (3) | 1 | 1 | 0 | 2 | 2 | 1
  Left Buttock (control): Extremely bothered (4) | 0 | 0 | 0 | 0 | 0 | 1
  Right Buttock: Extremely bothered (4) | 0 | 0 | 0 | 0 | 0 | 1

5. Secondary Outcome: Number of Participants With an Improved (+1 or Better) Score on the Investigator-Global Aesthetic Improvement Scale (I-GAIS) at Day 71
Description: Improvement was defined as +1 or better score on the I-GAIS for either buttock on Day 71 compared to Baseline. The I-GAIS is a 7-level scale ranging from +3 (very much improved) to -3 (very much worse). A higher score indicated a better outcome.
Time Frame: Day 71
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: CCH-aaes | Cohort 2: CCH-aaes + Compression Garment | Cohort 3: CCH-aaes + Instant Cold Packs | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) | Cohort 5: CCH-aaes + INhance Post-Injection Serum With TriHex Technology® | Cohort 6: CCH-aaes + PDL
Number analyzed (Participants) | 7 | 7 | 9 | 9 | 8 | 7
Participants
  Left Buttock (control) | 6 | 6 | 9 | 9 | 7 | 5
  Right Buttock | 6 | 6 | 9 | 9 | 7 | 6

6. Secondary Outcome: Number of Participants by Buttock at Each Level of Bruising on the Investigator Assessment of Bruising Severity Scale at Day 7
Description: Participants were assessed by the investigator using the Investigator Assessment of Bruising Severity Scale. The Investigator Assessment of Bruising Severity Scale is a 5-level scale ranging from 0 to 4, with "0" indicating no bruising or almost none, and "4" indicating very severe bruising. Higher scores indicated worse outcome.
Time Frame: Day 7
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: CCH-aaes | Cohort 2: CCH-aaes + Compression Garment | Cohort 3: CCH-aaes + Instant Cold Packs | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) | Cohort 5: CCH-aaes + Post-Injection Serum With TriHex Technology® | Cohort 6: CCH-aaes + PDL
Number analyzed (Participants) | 7 | 8 | 9 | 9 | 8 | 7
Participants
  Left Buttock (control): None or almost no bruising (0) | 0 | 0 | 0 | 0 | 0 | 1
  Right Buttock: None or almost no bruising (0) | 0 | 0 | 0 | 0 | 0 | 1
  Left Buttock (control): mild bruising (1) | 2 | 2 | 6 | 5 | 3 | 4
  Right Buttock: mild bruising (1) | 2 | 2 | 6 | 5 | 3 | 4
  Left Buttock (control): Moderate bruising (2) | 4 | 4 | 2 | 4 | 3 | 1
  Right Buttock: Moderate bruising (2) | 4 | 4 | 2 | 4 | 3 | 1
  Left Buttock (control): severe bruising (3) | 1 | 2 | 1 | 0 | 1 | 1
  Right Buttock: severe bruising (3) | 1 | 2 | 1 | 0 | 1 | 1
  Left Buttock (control): very severe bruising (4) | 0 | 0 | 0 | 0 | 1 | 0
  Right Buttock: severe bruising (4) | 0 | 0 | 0 | 0 | 1 | 0

7. Secondary Outcome: The Number of Participants by Buttock at Each Level of Bruising on the Investigator Assessment of Bruising Severity Scale at Day 14
Description: as for outcome 6
Time Frame: Day 14
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: CCH-aaes | Cohort 2: CCH-aaes + Compression Garment | Cohort 3: CCH-aaes + Instant Cold Packs | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) | Cohort 5: CCH-aaes + Post-Injection Serum With TriHex Technology® | Cohort 6: CCH-aaes + PDL
Number analyzed (Participants) | 7 | 7 | 9 | 9 | 8 | 7
Participants
  Left Buttock (control): None or almost no bruising (0) | 3 | 5 | 8 | 7 | 4 | 3
  Right Buttock: None or almost no bruising (0) | 3 | 6 | 9 | 8 | 4 | 3
  Left Buttock (control): mild bruising (1) | 4 | 2 | 1 | 2 | 2 | 4
  Right Buttock: mild bruising (1) | 4 | 1 | 0 | 1 | 4 | 4
  Left Buttock (control): Moderate bruising (2) | 0 | 0 | 0 | 0 | 2 | 0
  Right Buttock: Moderate bruising (2) | 0 | 0 | 0 | 0 | 0 | 0
  Left Buttock (control): severe bruising (3) | 0 | 0 | 0 | 0 | 0 | 0
  Right Buttock: severe bruising (3) | 0 | 0 | 0 | 0 | 0 | 0
  Left Buttock (control): very severe bruising (4) | 0 | 0 | 0 | 0 | 0 | 0
  Right Buttock: severe bruising (4) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: The Number of Participants by Buttock at Each Level of Bruising on the Investigator Assessment of Bruising Severity Scale at Day 22
Description: as for outcome 6
Time Frame: Day 22
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: CCH-aaes | Cohort 2: CCH-aaes + Compression Garment | Cohort 3: CCH-aaes + Instant Cold Packs | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) | Cohort 5: CCH-aaes + Post-Injection Serum With TriHex Technology® | Cohort 6: CCH-aaes + PDL
Number analyzed (Participants) | 6 | 7 | 9 | 9 | 8 | 7
Participants
  Left Buttock (control): None or almost no bruising (0) | 6 | 7 | 9 | 9 | 6 | 7
  Right Buttock: None or almost no bruising (0) | 6 | 7 | 9 | 9 | 7 | 7
  Left Buttock (control): mild bruising (1) | 0 | 0 | 0 | 0 | 2 | 0
  Right Buttock: mild bruising (1) | 0 | 0 | 0 | 0 | 1 | 0
  Left Buttock (control): Moderate bruising (2) | 0 | 0 | 0 | 0 | 0 | 0
  Right Buttock: Moderate bruising (2) | 0 | 0 | 0 | 0 | 0 | 0
  Left Buttock (control): severe bruising (3) | 0 | 0 | 0 | 0 | 0 | 0
  Right Buttock: severe bruising (3) | 0 | 0 | 0 | 0 | 0 | 0
  Left Buttock (control): very severe bruising (4) | 0 | 0 | 0 | 0 | 0 | 0
  Right Buttock: severe bruising (4) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Day 71
Groups:
- Cohort 3:CCH-aaes + Instant Cold Packs: CCH-aaes was administered to both buttocks with instant cold packs applied to the right buttock only for 5-10 minutes post injection as the mitigation treatment.
Arm/Group | Cohort 1: CCH-aaes | Cohort 2: CCH-aaes + Compression Garment | Cohort 3:CCH-aaes + Instant Cold Packs | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) | Cohort 5: CCH-aaes + INhance Post-Injection Serum With TriHex Technology® | Cohort 6: CCH-aaes + PDL
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/9 | 0/9 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/9 | 0/9 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 8/8 | 9/9 | 9/9 | 8/8 | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: CCH-aaes (N=7) | Cohort 2: CCH-aaes + Compression Garment (N=8) | Cohort 3:CCH-aaes + Instant Cold Packs (N=9) | Cohort 4: CCH-aaes + Arnica Gel Patches (OcuMend) (N=9) | Cohort 5: CCH-aaes + INhance Post-Injection Serum With TriHex Technology® (N=8) | Cohort 6: CCH-aaes + PDL (N=7)
Injection site bruising (General disorders) | 6 | 8 | 9 | 9 | 8 | 6
Injection site discolouration (General disorders) | 2 | 2 | 4 | 2 | 2 | 2
Injection site nodule (General disorders) | 1 | 2 | 2 | 0 | 0 | 3
Injection site pain (General disorders) | 4 | 5 | 7 | 7 | 5 | 5
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT04677712/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT04677712/SAP_001.pdf